CLINICAL TRIAL: NCT03705754
Title: EFFECT OF ENDOSCOPIC TATTOOING WITH CARBON BLACK SUSPENSION ON THE STAGING OF COLON CANCER
Brief Title: Carbon Black Tattoo in Colon Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Szeged University (Other)
Responsible Party: Principal Investigator, Matyas Czepan, Head of Division of Internal Medicine 2/S, Szeged University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/CCT
Record Dates: First submitted 2018-10-08; First posted 2018-10-15 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Endoscopic Tattoo of Suspected Colon Cancer

STUDY DESIGN:
Intervention Model Description: Tattoo arm vs. control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tattoo arm (Active Comparator): Tattoo will be placed by endoscopic submucosal injection of carbon black suspension
  Interventions: Device: carbon black suspension colonic tattoo injection
- Control arm (No Intervention): Tattoo will not be placed but case will follow standard procedure

INTERVENTIONS:
Device: carbon black suspension colonic tattoo injection — Examine the SPOT syringe to verify that the pigment is fully suspended. A 23 or 25 G sclerotherapy needle is recommended for this procedure, attach the syringe and prime with SPOT. After injection catheter is primed, manoeuver with the endoscope for optimal injection position and inject tangentially, at a 30-40˚ angle to the mucosa and create a saline bleb to find the submucosal plane prior to injecting SPOT to reduce risk of intramural injection. Document both the depth of scope and anatomic location of each tattoo and the ink consumption as well. Place injection 2-3 cm distal (downstream) of the area of interest. Use 0.5-0.75 mL per injection site and no more than 8 mL per patient. Place SPOT tattoos in 3-4 quadrants around the lumen to increase likelihood of visualisation.
  Other Names: GI supply SPOT endoscopic marker
  Arms: Tattoo arm

SUMMARY:
The study is designed to elucidate whether carbon black suspension endoscopic tattoo enhances visibility of lymph nodes or tumor tissue on dissection of colonic surgical specimen, thereby making improvement in staging defined as better pTNM stage via better visualisation of carbon marked metastatic or sentinel lymph nodes or marked primary tumor or adjacent tissues.

DETAILED DESCRIPTION:
Other objectives are:

* to assess intraoperative visibility of carbon black tattoo in the tumor region and surrounding tissues
* to assess microscopic distribution of carbon ink in the layers of the colonic wall and adjacent tissues
* to assess complications related to carbon black tattoo procedure like microscopic fibrosis, micro- or macroscopic scarring, inflammatory reactions
* to assess long-term effects of ink injections on control endoscopies at 6 and 12 months
* to assess dissection time in tattooed-non tattooed lymphatic tissues

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years or above undergoing colonoscopy for suspected colonic malignancy
* Participant is able to give informed consent for participation in the study
* Patient is presumably selected for surgery within 30 days following tattoo injection

Exclusion Criteria:

* Patients under the age of 18
* Patients unable to give informed consent or ineligible for surgery
* Tumor in the coecum dome or in the rectum (<15 cm)
* Known allergy to suspension ingredients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-02-06 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of tumors visualised from peritoneal cavity/number of tattoos visualised form peritoneal cavity | 1 year
  Distance in cm from tumor wich far carbon injection marked mucosa and adjacent tissues Number of inflammatory cells per field of view in injection site vs. non-injected mucosa Number of dissected total/normal/metastatic/carbon colored lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Matyas Czepan, MD, PhD, Principal Investigator — Szeged University
Locations (1):
- 1st Department of Medicine, University of Szeged, Szeged, Csongrád megye, Hungary

REFERENCES:
- [Result] Askin MP, Waye JD, Fiedler L, Harpaz N. Tattoo of colonic neoplasms in 113 patients with a new sterile carbon compound. Gastrointest Endosc. 2002 Sep;56(3):339-42. doi: 10.1016/s0016-5107(02)70035-7. PMID 12196769